CLINICAL TRIAL: NCT00134420
Title: Growth Hormone Trial for Children With 18q- and Abnormal Growth
Brief Title: Growth Hormone and Chromosome 18q- and Abnormal Growth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: South Texas Veterans Health Care System (U.S. Federal Agency); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 300-C07
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Loss of Chromosome 18q; Growth Hormone Deficiency
Keywords: Growth Hormone; Chromosomes, Human, Pair 18; Child
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone; Arginine; Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Growth Hormone Treatment (Active Comparator): Arginine and Clonidine Stimulation Testing, Growth Factors Laboratory Testing, and Neuropsychological Testing was done 1st for eligibility and this group received GH (growth hormone) (Nutropin AQ) 0.3 mgs per kg per week (standard dosing for GH)immediately after randomization
  Interventions: Drug: Nutropin AQ; Procedure: Arginine and Clonidine Stimulation Testing; Procedure: Growth Factors Laboratory Testing; Procedure: Neuropsychological Testing
- GH treatment delayed by one year (Other): Arginine and Clonidine Stimulation Testing, Growth Factors Laboratory Testing, and Neuropsychological Testing was done first for eligibility and this group received growth hormone (Nutropin AQ) 0.3 mgs per kg per week (standard dosing for GH)after one year of observation
  Interventions: Procedure: Arginine and Clonidine Stimulation Testing; Procedure: Growth Factors Laboratory Testing; Procedure: Neuropsychological Testing

INTERVENTIONS:
Drug: Nutropin AQ — Growth Hormone (Nutropin AQ) treatment given to Group 1 immediately Growth Hormone (Nutropin AQ) treatment given to Group 2 after one year observation
  Other Names: Growth Hormone (Nutropin AQ)
  Arms: Growth Hormone Treatment
Procedure: Arginine and Clonidine Stimulation Testing — This testing was done to determine growth hormone status prior to starting treatment.
Procedure: Growth Factors Laboratory Testing — This involved assessment of growth factors such as IGF#1 before treatment was initiated.
Procedure: Neuropsychological Testing — This testing was done prior to treatment and at the end of treatment.

SUMMARY:
We, the investigators at the University of Texas Health Science Center at San Antonio, want to learn if height and IQ (intelligence quotient) scores are improved by growth hormone (GH) treatment in children with chromosome 18 deletions and abnormal growth. Data from a previous study showed that growth hormone improved height in all children with 18q- and growth hormone deficiency. In addition, most of the study participants on growth hormone treatment showed an increase in IQ scores.

DETAILED DESCRIPTION:
HYPOTHESIS:

Our hypothesis with reference to children with 18q deletions who have abnormal growth are:

* growth hormone will improve growth; and
* growth hormone will improve performance IQ (pIQ).

Therefore, our specific aims are to evaluate the impact of GH treatment on:

* linear growth in children with 18q deletions who have abnormal growth but who are not classically growth hormone deficient; and
* pIQ in children with 18q deletions who have abnormal growth

GOALS AND METHODS:

We have already investigated the growth axis in 50 individuals with a cytogenetically and molecularly confirmed 18q deletion by determining the height, growth velocity, insulin-like growth factor 1 (IGF1), IGF binding protein 3 (IGFBP3), bone maturation and growth hormone (GH) response to pituitary stimulants (clonidine and arginine). To summarize: children with 18q deletions are short: 64% have a height more than 2 S.D. below the mean. Affected children also grow slowly: 68% have a growth velocity more than 1 S.D. below the mean. Half of the individuals have delayed bone maturation. Growth factors are skewed downward: 72% of the IGF1 values and 83% of the IGFBP3 values are below the average for normal children. Similarly, 72% of the children failed to adequately respond to the GH stimulants. In the total group of 50 children, 20 (40%) were classically GH DEFICIENT (height <-2 S.D., velocity <-1 S.D., bone age <-2 S.D., IGF1 < -1 S.D., IGFBP3 <-1 S.D., peak GH <10 ng/ml by polyclonal GH assay) and are on GH treatment. Of the remaining 30 children, 28 have multiple abnormalities of the growth axis, primarily growth velocity <-1 S.D. (ABNORMAL GROWTH), but did not qualify for GH treatment according to criteria set by their private insurer. Almost all of these children had abnormalities suggestive of hypothalamic dysfunction involving TSH (thyroid stimulating hormone) and prolactin. None have CNS (central nervous system) abnormalities of the pituitary on MRI. Thus we suspect that many of these children have neurosecretory dysfunction. Parental heights are slightly above average (father (height standard deviation score) HTZ = 0.3 +/- 1.2, mother HTZ = 0.1 +/- 1.1) and none of the children are overweight.

Of 8 children with GHD (growth hormone deficiency) on prolonged GH treatment, growth rates are comparable to those reported by the NCGS (National Collaborative Growth Study) for idiopathic GHD at 1 and 2 years. The mean change in height over a 28-month period for the treated group in our study was +1.8 S.D. while it was -0.25 S.D. in the untreated group (p<0.001). No known complications of GH treatment were encountered. Furthermore, because of an association between 18q deletion, hypomyelination and cognition, some non-statural benefits of GH treatment were examined: specifically, the performance intelligence quotient (pIQ) was measured using a detailed battery of neuropsychological instruments. The pIQ was measured because many of the children are hearing impaired and a full scale IQ, which relies on verbal skills, would underestimate their abilities. The GH-treated group was compared to an untreated group. The GH-treated group (n=8) showed an increase in pIQ of 23 points (range 0 to +47) while the untreated group (n=6) showed no change (range -2 to +6)(p=0.003). Based on these observations, we conclude that GHD children with 18q deletions respond favorably to GH therapy in terms of both linear growth and pIQ. In contrast, children with 18q deletions with abnormal growth who are not classically GH deficient, show little change in height S.D. and pIQ over time. Therefore, we propose to study (NEW STUDY) whether children with 18q deletions with abnormal growth can benefit from GH treatment. For purposes of this proposal, abnormal growth is defined as a growth velocity <-1 S.D.

Initial auxology, endocrine testing, and neurocognitive evaluation will be performed at our Center. Auxologic and neurocognitive testing will be repeated after 18 months of therapy at our Center. These studies are done at our Center to assure consistency of evaluation, which is a particular concern for the neurocognitive tests. Many of the children will also participate in other studies in our Center (MRI imaging, psychological evaluations of family function) that are not part of this application. Children begun on GH treatment will need to be seen by a pediatric endocrinologist for dosage adjustment after 3, 6, 9 and 12 months. The untreated children will also need to be seen by a pediatric endocrinologist for auxologic studies at the same time points. We enrolled 20 children in this study. Few of the children are located in any single geographic area; therefore, we will have 12-20 centers seeing individual children. Rather than developing new forms, standard NCGS intake forms will be used for the intermediate visits by the local pediatric endocrinologists.

Control Group: We have more than 20 previously studied children, 5.3 +/- 2.8 years of age, who have abnormal growth and have never received GH. All have undergone extensive auxologic, hormonal, neurocognitive and neuroimaging evaluations. These studies were done 15.4 +/- 9 months ago (range 11-28 months). We have already shown that, in the absence of intervention, height S.D. and pIQ are stable over time; therefore, these children can serve as their own controls.

We also have 20 children who are GH deficient and on treatment that are participants in another study. These children were evaluated prior to the initiation of treatment. All are scheduled to be re-evaluated at least twice in a five-year period. The data on the first 8 treated children were reported above. These children will serve as important "disease controls".

NAME OF FDA APPROVED DRUG TO BE USED:

We are using Nutropin AQ in this study.

METHOD OF TREATMENT ASSIGNMENT:

All children who have previously been evaluated in our Center were offered the opportunity to receive GH, subject to the following limitations:

* The prior evaluation must have occured at least 12 months preceding the anticipated date of initiation of GH therapy.
* May not be on GH treatment or have been previously treated with GH
* Growth velocity <-1 S.D. with normal weight for length/height
* Must be willing to return to our Center for reevaluation of auxologic parameters and neurocognitive testing prior to the initiation of GH therapy.
* Must be willing to administer GH on a daily basis for 12-15 months
* Must be willing to return to our Center for re-evaluation after 12-15 months of therapy.

The majority of the 20 patients for this study came from the group of children who have been previously evaluated.

New children (families) being seen for their initial visit in our Center, will be offered the opportunity to participate in the clinical trial if they have abnormal growth and are not classically GHD. However, these children will be randomly assigned either to treatment or non-treatment for the initial 12-month period. Both treated and untreated children (families) must comply with limitations 2-6 above.

The minority of the 20 patients for this study came from the group of children who are new.

TYPE OF RANDOMIZATION:

Randomization applied only to children who are new to our Center. When the results of growth factor and GH provocative testing are known, a two-step process will occur. Children, who are GHD, will be started on GH and entered into an on-going study already underway in our Center. They will not qualify for participation in the proposed NEW study. Children who have abnormal growth will be assigned to either the treatment or non-treatment category, using an adaptive randomization scheme to avoid imbalances in the numbers of subjects allocated to the two groups.

PLANNED INTERIM ANALYSIS:

GH-treated children will be seen at 3, 6, 9 and 12 months by their local pediatric endocrinologist for measurement of height and weight, review of medical history and dosage adjustment. Untreated children will be seen at 3, 6, 9, and 12 months for measurement of height and weight and review of medical history.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chromosome 18 deletion (cytogenetics report)
* Children with abnormal growth but who are not classically growth hormone deficient

Exclusion Criteria:

* Children previously on growth hormone therapy

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2001-02; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
growth rates 12-15 months after treatment begins

SECONDARY OUTCOMES:
performance IQ scores 12-15 months after treatment begins

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E. Hale, M.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States